CLINICAL TRIAL: NCT05045313
Title: A Three-part, Single-center, Open-label, Phase I Clinical Study to Evaluate the Drug-drug Interactions (DDIs) Between DBPR108 and Warfarin Sodium/Digoxin/Probenecid in Healthy Subjects
Brief Title: A Study to Evaluate the Drug-drug Interactions (DDIs) of DBPR108 With Warfarin Sodium, Digoxin, Probenecid in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA1118-CSP-012
Record Dates: First submitted 2021-08-05; First posted 2021-09-16 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-08

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Warfarin; Digoxin; Probenecid; DBPR108

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The DDI of DBPR108 and Warfarin Sodium Tablets (Experimental): Subjects will receive a single dose of Warfarin sodium 5 mg on Day 1, then take DBPR108 100 mg once-daily on Day 15 through Day 26 and a single dose of Warfarin sodium 5 mg on Day 19.
  Interventions: Drug: Warfarin sodium tablets; Drug: DBPR108 tablets
- The DDI of DBPR108 and Digoxin Tablets (Experimental): Subjects will receive a single dose of Digoxin 0.25 mg on Day 1, then take DBPR108 100 mg once-daily on Day 6 through Day 15 and a single dose of Digoxin 0.25 mg on Day 10.
  Interventions: Drug: Digoxin tablet; Drug: DBPR108 tablets
- The DDI of DBPR108 and Probenecid Tablets (Experimental): Subjects will receive a single dose of DBPR108 100 mg on Day 1, then take Probenecid 500 mg twice-daily on Day 5 through Day 9 and a single dose of DBPR108 100 mg on Day 7.
  Interventions: Drug: Probenecid tablets; Drug: DBPR108 tablets

INTERVENTIONS:
Drug: Warfarin sodium tablets — Drug: Warfarin sodium, tablet, oral
  Arms: The DDI of DBPR108 and Warfarin Sodium Tablets
Drug: Digoxin tablet — Drug: Digoxin, tablet, oral
  Arms: The DDI of DBPR108 and Digoxin Tablets
Drug: Probenecid tablets — Drug: Probenecid, tablet, oral
  Arms: The DDI of DBPR108 and Probenecid Tablets
Drug: DBPR108 tablets — Drug: DBPR108, tablet, oral
  Other Names: DBPR108

SUMMARY:
This is a three-part, single-center, open-label phase I clinical study to characterize the DDIs potential of DBPR108 with Warfarin sodium, Digoxin, or Probenecid in healthy subjects. This study also aims to evaluate the safety and tolerability of DBPR108 in the presence of Warfarin sodium, Digoxin, or Probenecid.

DETAILED DESCRIPTION:
DBPR108 is a potent dipeptidylpeptidase-4 inhibitor. This study will be run in three parts to characterize the DDIs potential of DBPR108 with the expected concomitant drugs (Warfarin sodium, Digoxin, Probenecid) in Healthy Subjects. Each part of this study consists of a screening period (Day -14 to Day -1), a baseline period (Day -1), a treatment period, and a follow-up visit period. Approximately 14 subjects will be enrolled in each part of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions;
2. 18 to 45 years (inclusive), male and female;
3. Male subjects weight ≥50.0 kg and female subjects weight ≥45.0 kg. Body mass index (BMI): 18-28 kg/m^2 (inclusive) (BMI= weight (kg)/height^2 (m^2)；
4. Subjects (including their partners) are willing to use effective contraceptives from screening to the 6 months after the last dose administration;
5. Subjects judged to be in good health by the investigator, based on the physical examination, vital signs examination, 12-lead electrocardiogram (ECG) examination and laboratory examination etc;

Exclusion Criteria:

1. Subjects who have a history of allergic conditions (such as asthma, urticaria), or have a history of allergy to any of the study drugs or other similarly structured drugs;
2. Subjects with a history of severe diseases, such as cardiovascular, respiratory, liver, gastrointestinal, endocrine, hematological, psychiatric/neurological systems diseases within 1 year prior to screening;
3. Subjects with a history of hypoglycemia or abnormal blood glucose at screening: fasting blood glucose <70 mg/dL (3.9 mmol/L) or >110 mg/dL (6.1 mmol/L);
4. Subjects who have previously undergone surgery that may affect the absorption, distribution, metabolism, or excretion of the drug (e.g., subtotal gastrectomy), or who have a scheduled surgical plan during the study period;
5. Use of any prescription drug, over-the-counter drug, or herbal medicine within 2 weeks prior to screening;
6. Have been vaccinated within 4 weeks prior to screening or who have a scheduled vaccinated plan during the study period;
7. History of drug abuse, or positive urine drug screen at screening;
8. Smoking more than 5 cigarettes per day within 3 months prior to screening，or who cannot stop using any tobacco products during the study period；
9. Average daily intake of alcohol is more than 28 g alcohol (male) or 14 g (female) (14 g ≈ 497 mL beer, or 44 mL spirits with low alcohol content, or 145 mL wine) within the 3 months prior to screening, or taking any product containing alcohol within 48 h before dosing, or a positive ethanol breath test at screening;
10. Consumption of grapefruit juice, methylxanthine-rich food or beverage (such as coffee, tea, cola, chocolate, energy drinks) within 48 h before the administration, or those who have had strenuous exercise, or have other factors affecting drug absorption, distribution, metabolism, excretion, etc;
11. Participation in another clinical trial within 3 months before screening (whichever is administrated)；
12. Blood donation (or blood loss) ≥400 mL, or receiving whole blood transfusions or erythrocyte suspension transfusions within 3 months prior to the screening;
13. Any positive test result of hepatitis B surface antigen, hepatitis C virus antibody, anti-human immunodeficiency virus antibody or anti-Treponema pallidum specific antibody;
14. Pregnant/lactating woman, or has a positive pregnancy test at screening;
15. Not suitable for this study as judged by the investigator;
16. Supplementary exclusion criteria for the first part of the study: subjects with bleeding tendency, or PT and INR test results judged by the investigator to be not suitable for participating in the study;
17. Supplementary exclusion criteria for the third part of the study: the estimated glomerular filtration rate (eGFR) calculated by the modification of diet in renal diseases (MDRD) equation at screening with clinical significance as judged by the investigator, or subjects with nephrolithiasis or have a history of nephrolithiasis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Part one: Peak plasma concentration (Cmax) of S-warfarin and R-warfarin | Day 1 to Day 8, and Day 19 to Day 26
Part one: Area under the plasma concentration versus time curve (AUC) of S-warfarin and R-warfarin | Day 1 to Day 8, and Day 19 to Day 26
Part one: Peak plasma concentration (Cmax) of DBPR108 | Day 17 to Day 20
Part one: Area under the plasma concentration versus time curve (AUC) of DBPR108 | Day 17 to Day 20
Part two: Peak plasma concentration (Cmax) of Digoxin | Day 1 to Day 6, and Day 10 to Day 15
Part two: Area under the plasma concentration versus time curve (AUC) of Digoxin | Day 1 to Day 6, and Day 10 to Day 15
Part two: Peak plasma concentration (Cmax) of DBPR108 | Day 8 to Day 11
Part two: Area under the plasma concentration versus time curve (AUC) of DBPR108 | Day 8 to Day 11
Part three: Peak plasma concentration (Cmax) of DBPR108 | Day 1 to Day 3, and Day 7 to Day 9
Part three: Area under the plasma concentration versus time curve (AUC) of DBPR108 | Day 1 to Day 3, and Day 7 to Day 9

SECONDARY OUTCOMES:
Part one: Time to achieve maximum plasma concentration (Tmax) of S-warfarin and R-warfarin | Day 1 to Day 8, and Day 19 to Day 26
Part one: Half-life(t1/2) of S-warfarin and R-warfarin | Day 1 to Day 8, and Day 19 to Day 26
Part one: Apparent volume of Distribution(Vz/F) of S-warfarin and R-warfarin | Day 1 to Day 8, and Day 19 to Day 26
Part one: Apparent clearance(CL/F) of S-warfarin and R-warfarin | Day 1 to Day 8, and Day 19 to Day 26
Part one: Time to achieve maximum plasma concentration (Tmax) of DBPR108 | Day 17 to Day 20
Part one: Half-life(t1/2) of DBPR108 | Day 17 to Day 20
Part one: Apparent volume of Distribution(Vz/F) of DBPR108 | Day 17 to Day 20
Part one: Apparent clearance(CL/F) of DBPR108 | Day 17 to Day 20
Part one: the pharmacodynamic parameters-Prothrombin time(PT) | Day 1 to Day 8, and Day 19 to Day 26
Part one: the pharmacodynamic parameters-International normalized ratio(INR) | Day 1 to Day 8, and Day 19 to Day 26
Part two: Time to achieve maximum plasma concentration (Tmax) of Digoxin | Day 1 to Day 6, and Day 10 to Day 15
Part two: Half-life(t1/2) of Digoxin | Day 1 to Day 6, and Day 10 to Day 15
Part two: Apparent volume of Distribution(Vz/F) of Digoxin | Day 1 to Day 6, and Day 10 to Day 15
Part two: Apparent clearance(CL/F) of Digoxin | Day 1 to Day 6, and Day 10 to Day 15
Part two: Time to achieve maximum plasma concentration (Tmax) of DBPR108 | Day 8 to Day 11
Part two: Half-life(t1/2) of DBPR108 | Day 8 to Day 11
Part two: Apparent volume of Distribution(Vz/F) of DBPR108 | Day 8 to Day 11
Part two: Apparent clearance(CL/F) of DBPR108 | Day 8 to Day 11
Part three: Time to achieve maximum plasma concentration (Tmax) of DBPR108 | Day 1 to Day 3, and Day 7 to Day 9
Part three: Half-life(t1/2) of DBPR108 | Day 1 to Day 3, and Day 7 to Day 9
Part three: Apparent volume of Distribution(Vz/F) of DBPR108 | Day 1 to Day 3, and Day 7 to Day 9
Part three: Apparent clearance(CL/F) of DBPR108 | Day 1 to Day 3, and Day 7 to Day 9
Part three:Cumulative amount of drug excreted in urine(Ae) of DBPR108 | Day 1 to Day 3, and Day 7 to Day 9
Part three: Cumulative fraction of the dose excreted(fe) of DBPR108 | Day 1 to Day 3, and Day 7 to Day 9
Part three: Renal Clearance(CLR) of DBPR108 | Day 1 to Day 3, and Day 7 to Day 9
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Number of participants with treatment-related adverse events will be assessed by CTCAE v5.0. The AEs will be summarized according to the system organ class (SOC) and preferred term (PT), including the number and percentage of participants who had AEs.
Clinically significant changes from baseline in 12-lead electrocardiogram (ECG) examination will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  ECG monitoring includes heart rate in bpm.
Clinically significant changes from baseline in 12-lead electrocardiogram (ECG) examination will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  ECG monitoring includes P-R, QT and QTc intervals in ms.
Clinically significant changes from baseline in physical examination will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Physical examination includes general conditions, skin, mucous membranes, head, neck, chest, abdomen, spine, limbs, nervous system, and lymphatic system.
Clinically significant changes from baseline in vital signs examination will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Vital signs monitoring includes body temperature in degrees Celsius.
Clinically significant changes from baseline in vital signs examination will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Vital signs monitoring includes respiratory rate and pulse in times per minute.
Clinically significant changes from baseline in vital signs examination will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Vital signs monitoring includes systolic blood pressure and diastolic blood pressure in mmHg.
Clinically significant changes from baseline in routine blood test will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Routine blood test includes red blood cell count in 10^12/L.
Clinically significant changes from baseline in routine blood test will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Routine blood test includes hemoglobin in g/L.
Clinically significant changes from baseline in routine blood test will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Routine blood test includes hematocrit in L/L.
Clinically significant changes from baseline in routine blood test will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Routine blood test includes white blood cell count, platelet, neutrophilic granulocyte count, lymphocyte count and monocyte count in 10^9 /L.
Clinically significant changes from baseline in blood biochemistry test will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Blood biochemistry test includes total protein and albumin in g/L.
Clinically significant changes from baseline in blood biochemistry test will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Blood biochemistry test includes alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase and glutamyltranspeptidase in U/L.
Clinically significant changes from baseline in blood biochemistry test will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Blood biochemistry test includes total bilirubin and serum creatinine in umol/L.
Clinically significant changes from baseline in blood biochemistry test will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Blood biochemistry test includes urea in mmol/L.
Clinically significant changes from baseline in routine urine test will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Routine urine test includes urobilinogen, glucose and protein in mg/dL.
Clinically significant changes from baseline in routine urine test will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Routine urine test includes pH.
Clinically significant changes from baseline in coagulation function test will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Coagulation action test includes fibrinogen in g/L.
Clinically significant changes from baseline in coagulation function test will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Coagulation action test includes prothrombin time, thrombin time and activated partial thromboplatin time in seconds.
Clinically significant changes from baseline in coagulation function test will be recorded as AEs at each visit time point. | Up to Day 33 from screening for part one, up to Day 22 from screening for part two, and up to Day 16 from screening for part three.
  Coagulation action test includes international normalized ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, China